CLINICAL TRIAL: NCT04685798
Title: Optimized Diffusion-Weighted Imaging for the Evaluation of Post-Treatment Squamous Cell Carcinoma in the Neck: Comparative Study With FDG PET/CT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201912072
Record Dates: First submitted 2020-11-24; First posted 2020-12-28 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Diffusion Magnetic Resonance Imaging

STUDY DESIGN:
Masking Description: All anonymized MRI studies will be blindly evaluated by at least two experienced neuroradiologists
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- DWI MRI + Standard of care FDG PET/CT (Experimental): -The patients will undergo an optimized research neck DWI MRI, up to 3 weeks post-treatment and then a standard-of-care 3-month post-treatment FDG PET/CT examination.
  Interventions: Device: Diffusion-weighted imaging magnetic resonance imaging; Device: FDG PET/CT

INTERVENTIONS:
Device: Diffusion-weighted imaging magnetic resonance imaging — The research MRI study of the head and neck will be performed on a Siemens 3T MRI Scanner system
  Other Names: DWI MRI
Device: FDG PET/CT — Standard of care

SUMMARY:
The investigators propose a longitudinal study evaluating post-treatment changes in patients with squamous cell carcinoma (SCC) of the neck using an innovative optimized diffusion-weighted imaging (DWI) pulse sequence to identify more accurately recurrent tumors as well as early non-responders to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven newly diagnosis or recurrence as indicated by tissue diagnosis of T3 or T4 squamous cell carcinoma of the head and neck
* Must have had or be scheduled for standard-of-care surgical resection, radiation, and/or chemo-radiation of the diagnosed squamous cell carcinoma of the head and neck
* At least 18 years of age
* Patient must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Contraindications to MRI, including:

  * MRI-incompatible implantable devices
  * severe claustrophobia; and
* Pregnant and/or breastfeeding, with women of childbearing potential having a negative urine or serum pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria J Guzman Pérez-Carrillo, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DWI MRI + Standard of Care FDG PET/CT
Started | 8
Completed | 6
Not Completed | 2
Not completed — Did not have standard of care FDG PET/CT | 2

BASELINE CHARACTERISTICS:
Arm/Group | DWI MRI + Standard of Care FDG PET/CT
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: years] | 61 [42 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Apparent Diffusion Coefficient Mean (ADCmean)
Description: * ADC=measure of the magnitude of diffusion (of water molecules) within tissue
  * The primary tumor, suspicious lesion, and/or area of post-treatment change will be identified in anatomical images & then outlined in the ADC sequence, excluding areas of cystic change and necrosis. If there are multiple lesions, only the dominant lesion with the lowest ADC will be used for analysis
  * A histogram analysis method will examine the distribution of ADC values within each region of interest (ROI)
  * ADCmean will describe distribution of ADC measurements in tumor/non-tumor tissues & independent sample t-test will compare ADC measurements between the 2 groups
Time Frame: 2-3 weeks post-standard of care treatment
Population: Evaluable patients include those that received the DWI MRI and the standard of care FDG PET/CT, had measurable disease on imaging, and had tumor persistence/recurrence.
Measure: Mean (Standard Deviation); unit: x 10-6 mm^2/s
Arm/Group | DWI MRI + Standard of Care FDG PET/CT
Number analyzed (Participants) | 1
x 10-6 mm^2/s | 1.337 (NA) — There is only participant evaluable.

2. Primary Outcome: Apparent Diffusion Coefficient Lowest Value in a Tumor (ADCmin)
Description: * ADC=measure of the magnitude of diffusion (of water molecules) within tissue
  * The primary tumor, suspicious lesion, and/or area of post-treatment change will be identified in anatomical images & then outlined in the ADC sequence, excluding areas of cystic change and necrosis. If there are multiple lesions, only the dominant lesion with the lowest ADC will be used for analysis
  * A histogram analysis method will examine the distribution of ADC values within each region of interest (ROI)
  * ADCmin will describe distribution of ADC measurements in tumor/non-tumor tissues & independent sample t-test will compare ADC measurements between the 2 groups
Time Frame: 2-3 weeks post-standard of care treatment
Population: as for outcome 1
Measure: Number; unit: x 10-6 mm^2/s
Arm/Group | DWI MRI + Standard of Care FDG PET/CT
Number analyzed (Participants) | 1
x 10-6 mm^2/s | 1.007

3. Secondary Outcome: Number of Participants That Were Non-responders to Treatment on Both the DWI MRI and the Standard of Care FDG PET/CT
Time Frame: 2-3 weeks post-standard of care treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | DWI MRI + Standard of Care FDG PET/CT
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of MRI through completion of MRI (approximately 3 hours). Adverse events were not collected for the standard of care FDG PET/CT.
Arm/Group | DWI MRI + Standard of Care FDG PET/CT
All-Cause Mortality (participants affected / at risk) | 3/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/98/NCT04685798/Prot_SAP_000.pdf